CLINICAL TRIAL: NCT04554459
Title: Ponatinib Plus Reduced-intensity Chemotherapy in the First-line Treatment of Adult Patients With Ph-positive Acute Lymphoblastic Leukemia
Brief Title: Ponatinib Plus Reduced-intensity Chemotherapy in the First-line Treatment of Adult Patients With Ph+ ALL
Acronym: Pona-CELL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slower recruitment rate;
Sponsor: Institute of Hematology and Blood Transfusion, Czech Republic (Other)
Collaborators: CZECRIN - Czech Clinical Research Infrastructure Network (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pona-CELL
Record Dates: First submitted 2020-09-04; First posted 2020-09-18 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2023-08

CONDITIONS: Acute Lymphoblastic Leukemia, Adult; Ph+ ALL; Newly Diagnosed
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — ponatinib; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ponatinib plus reduced-intensity chemotherapy (Experimental): ponatinib plus reduced-intensity chemotherapy in first-line treatment of Adult Ph+ ALL
  Interventions: Drug: Ponatinib 15 MG Oral Tablet

INTERVENTIONS:
Drug: Ponatinib 15 MG Oral Tablet — ponatinib plus reduced-intensity chemotherapy in first-line treatment of Adult Ph+ ALL
  Other Names: Iclusig; AP24534; L01XE24

SUMMARY:
This is a phase II interventional trial to evaluate the efficacy of ponatinib plus reduced-intensity chemotherapy in the first-line treatment of adult patients with Ph+ acute lymphoblastic leukemia. This combination has the potential to improve the depth of molecular responses after the induction phase of treatment. Patients who achieve a complete molecular response (CMR) at week 11 will not be directed to alloSCT and will receive consolidation chemotherapy combined with ponatinib, followed by 24 months of ponatinib maintenance. The aim is to spare individuals with a low probability of relapse from overtreatment with more intensive and toxic transplant procedure.

DETAILED DESCRIPTION:
Primary Objective:

To evaluate the percentage of complete molecular responses (CMR) after two cycles of remission induction therapy composed of two cycles of chemotherapy plus ponatinib. CMR is defined as BCR-ABL1 below the Limit of Quantification by Droplet Digital Polymerase Chain Reaction (ddPCR).

Outline:

Pre-phase:

dexamethasone 10 mg/m2 PO (day -5 till -1), cyclophosphamide IV 200 mg/m2 (day -3 till -1), methotrexate 15 mg IT.

Induction I:

ponatinib 30 mg/day PO once daily (QD) continuously since day 1, rituximab 375 mg/m2 IV (day 1), dexamethasone 10 mg/m2 PO (day 1-2, 8-11), vincristine 2 mg IV (day 1, 8, 15), Granulocyte-Colony Stimulating Factor (G-CSF) until recovery.

Induction II:

ponatinib 30 mg/day PO QD continuously, rituximab 375 mg/m2 IV (day 23), cyclophosphamide 1000 mg/m2 IV (day 24), cytarabine 75 mg/m2 IV (day 26-29, 33-36), Granulocyte StimuG-CSF until recovery, methotrexate 15 mg IT (day 26, 33) methotrexate 15 mg + cytarabine 40 mg + dexamethasone 4 mg IT (day 40). Week 11: Primary endpoint assessment.

Consolidation I (week 12):

ponatinib 30 mg/day PO QD continuously, rituximab 375 mg/m2 IV (day 1), dexamethasone 10 mg/m2 PO (day 1-4), vindesine 3 mg/m2 IV (day 2), methotrexate 1.5 g/m2 IV (day 2), cytarabine 2x 2 g/m2 IV (day 5), G-CSF until recovery, methotrexate 15 mg + cytarabine 40 mg + dexamethasone 4 mg IT (day 8). Patients in complete molecular response at week 11 will be treated with 5 additional blocks of chemotherapy followed by maintenance therapy; patients with molecular failure at week 11 will end the study and be directed to alloSCT.

Consolidation II (week 18):

ponatinib 15 mg/day PO QD continuously, rituximab 375 mg/m2 IV (day 1), cyclophosphamide 500 mg/m2 IV (day 2,3), etoposide (VP-16) 75 mg/m2 IV (day 2,3), methotrexate 15 mg + cytarabine 40 mg + dexamethasone 4 mg IT (day 1).

Consolidation III+V (weeks 24 and 36):

ponatinib 15 mg/day PO QD continuously, rituximab 375 mg/m2 IV (day 1), methotrexate 1.5 g/m2 IV (day 2), vincristine 1 mg IV (day 2), 6-mercaptopurine 60 mg/m2 PO (day 2-8), methotrexate 15 mg + cytarabine 40 mg + dexamethasone 4 mg IT at day 1.

Consolidation IV+VI (weeks 30+40):

ponatinib 15 mg/day PO QD continuously, rituximab 375 mg/m2 IV (day 1), dexamethasone 10 mg/m2 PO (day 1-4), cytarabine 1.5 g/m2 IV (day 1+3+5), methotrexate 15 mg + cytarabine 40 mg + dexamethasone 4 mg IT (day 1). Maintenance: ponatinib 15 mg/day PO QD continuously 24 months. (Doses of IV methotrexate and cytarabine are reduced in patients >55 years.)

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed, previously untreated, Ph-positive [either t(9;22) and/or BCR-ABL positive] B-precursor acute lymphoblastic leukemia;
* Age more than 18 years;
* Eligible to intensive chemotherapy, due to general health status;
* ECOG (Eastern Cooperative Oncology Group) performance status ≤2;
* Absence of significant liver disease, as defined by the following criteria: total serum bilirubin ≤1.5 x upper limit of normal (ULN), unless due to Gilbert's syndrome, alanine aminotransferase (ALT) ≤2.5 × ULN or ≤5 x ULN if leukemic involvement of the liver is present, and aspartate aminotransferase (AST) ≤2.5 × ULN or ≤5 x ULN if leukemic involvement of the liver is present;
* Adequate pancreatic function as defined by serum amylase and lipase ≤1.5 × ULN;
* Diagnostic sample of bone marrow (or peripheral blood with >50% of blasts) available for central MRD assessment;
* Subject has provided written informed consent prior to any screening procedure.

Exclusion Criteria:

* Lymphoid blast crisis of chronic myelocytic leukemia (CML);
* Active serious infection not controlled by oral or intravenous antibiotics;
* Active known hepatitis B virus (HBV) or hepatitis C virus (HCV) or positive HIV serology;
* History of acute pancreatitis within 1 year of study or history of chronic pancreatitis;
* Uncontrolled hypertriglyceridemia (triglycerides > 5.1 µmol/L);
* Clinically significant, uncontrolled or active cardiovascular disease, specifically including, but not restricted to: any history of myocardial infarction, stroke, or revascularization; unstable angina or transient ischemic attack within 6 months prior to enrolment; congestive heart failure within 6 months prior to enrolment or left ventricular ejection fraction (LVEF) less than lower limit of normal per local institutional standards; history of clinically significant (as determined by the treating physician) atrial arrhythmia; any history of ventricular arrhythmia; any history of venous thromboembolism including deep venous thrombosis or pulmonary embolism;
* Uncontrolled hypertension (diastolic blood pressure >90 mmHg; systolic >140 mmHg). Patients with hypertension should be under treatment on study entry to effect blood pressure control;
* Creatinine levels > 160 µmol/L or estimated creatinine clearance of < 50 mL/min;
* GI disease and/or major GI surgery that may significantly alter the absorption of study drug
* Hypersensitivity to the active substance or to any of the excipients, especially galactose intolerance.
* Taking any medications or herbal supplements that are known to be strong inhibitors of CYP3A4 within at least 14 days before the first dose of ponatinib;
* Female patients who are pregnant or breast feeding or patients of childbearing potential not willing to use a highly effective method of contraception during the study and for 3 months following the last dose of study drug;
* Male patients whose sexual partner(s) are women of childbearing potential who are not willing to use a highly effective method of contraception, one of which includes a condom, during the study;
* Patients with a history of another primary malignancy that is currently clinically significant or currently requires active intervention;
* Any concurrent severe and/or uncontrolled medical condition, which could, in the opinion of the investigator, compromise participation in the study;
* Concurrent participation in another clinical study with an investigational medical product.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Complete Molecular Response | At week 11 (acceptable window + 1 wk); after completion of two induction courses and before starting of the 1st Consolidation cycle (each induction course is 23 days with continuing ponatinib treatment till the outcome assessing)
  Percentage of patients with Complete Molecular Response (CMR) after 2 cycles of induction therapy composed by reduced chemotherapy and ponatinib. Minimal Residual Disease (MRD) tested by quantification of BCR-ABL1 transcript using ddPCR method

SECONDARY OUTCOMES:
CR and CRi | CR and CRi at the end of the 1st Induction Course (Day 23) and at week 11 (acceptable window + 1wk) after completion of the 2nd Induction Course and before starting of the 1st Consolidation Cycle
  Complete Remission (CR) and Complete Remission with incomplete blood count recovery(CRi)
PFS | Time from the day of CR/CRi documentation until the date of relapse, or death from any cause whichever came first, assessed up to 36 months
  Progression Free Survival (PFS)
OS | Time from the day 1 (starting of the 1st Induction Course) until the date of death from any cause, assessed up to 36 months
  Overall Survival (OS)
AlloSCT in the first complete remission | At week 11 (acceptable window + 1 wk); after completion of two induction courses and before starting of the 1st Consolidation cycle (each induction course is 23 days with continuing ponatinib treatment till the outcome assessing)
  Percentage of patients with suboptimal molecular response after completion of 2 induction course containing ponatinib
Severity and occurence of adverse events related to ponatinib | During the ponatinib treatment up to 30 days after end of treatment
  Severity and occurence of adverse events related to ponatinib treatment

CONTACTS AND LOCATIONS:
Overall Officials: Cyril Salek, MD, Principal Investigator — Institute of Hematology and Blood Transfusion, Czech Republic
Locations (7):
- Czechia (7):
  - University Hospital Brno, Internal hematology and oncology clinic, Brno
  - University Hospital Hradec Kralove, The 4th Department of Internal Medicine - Hematology, Hradec Králové
  - University Hospital Olomouc, Hematooncology Clinic, Olomouc
  - University Hospital Ostrava, Hematooncology Clinic, Ostrava
  - University Hospital Plzen, Hematology and Oncology Department, Plzeň-Lochotín
  - University Hospital Kralovske Vinohrady, Internal Hematology Clinic, Prague
  - Institute of Hematology and Blood Transfusion, Prague

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Daver N, Thomas D, Ravandi F, Cortes J, Garris R, Jabbour E, Garcia-Manero G, Borthakur G, Kadia T, Rytting M, Konopleva M, Kantarjian H, O'Brien S. Final report of a phase II study of imatinib mesylate with hyper-CVAD for the front-line treatment of adult patients with Philadelphia chromosome-positive acute lymphoblastic leukemia. Haematologica. 2015 May;100(5):653-61. doi: 10.3324/haematol.2014.118588. Epub 2015 Feb 14. PMID 25682595
- [Background] Bassan R, Rossi G, Pogliani EM, Di Bona E, Angelucci E, Cavattoni I, Lambertenghi-Deliliers G, Mannelli F, Levis A, Ciceri F, Mattei D, Borlenghi E, Terruzzi E, Borghero C, Romani C, Spinelli O, Tosi M, Oldani E, Intermesoli T, Rambaldi A. Chemotherapy-phased imatinib pulses improve long-term outcome of adult patients with Philadelphia chromosome-positive acute lymphoblastic leukemia: Northern Italy Leukemia Group protocol 09/00. J Clin Oncol. 2010 Aug 1;28(22):3644-52. doi: 10.1200/JCO.2010.28.1287. Epub 2010 Jul 6. PMID 20606084
- [Background] Bruggemann M, Raff T, Kneba M. Has MRD monitoring superseded other prognostic factors in adult ALL? Blood. 2012 Nov 29;120(23):4470-81. doi: 10.1182/blood-2012-06-379040. Epub 2012 Oct 2. PMID 23033265
- [Background] Cortes JE, Kim DW, Pinilla-Ibarz J, le Coutre P, Paquette R, Chuah C, Nicolini FE, Apperley JF, Khoury HJ, Talpaz M, DiPersio J, DeAngelo DJ, Abruzzese E, Rea D, Baccarani M, Muller MC, Gambacorti-Passerini C, Wong S, Lustgarten S, Rivera VM, Clackson T, Turner CD, Haluska FG, Guilhot F, Deininger MW, Hochhaus A, Hughes T, Goldman JM, Shah NP, Kantarjian H; PACE Investigators. A phase 2 trial of ponatinib in Philadelphia chromosome-positive leukemias. N Engl J Med. 2013 Nov 7;369(19):1783-96. doi: 10.1056/NEJMoa1306494. Epub 2013 Nov 1. PMID 24180494
- [Background] DeBoer R, Koval G, Mulkey F, Wetzler M, Devine S, Marcucci G, Stone RM, Larson RA, Bloomfield CD, Geyer S, Mullighan CG, Stock W. Clinical impact of ABL1 kinase domain mutations and IKZF1 deletion in adults under age 60 with Philadelphia chromosome-positive (Ph+) acute lymphoblastic leukemia (ALL): molecular analysis of CALGB (Alliance) 10001 and 9665. Leuk Lymphoma. 2016 Oct;57(10):2298-306. doi: 10.3109/10428194.2016.1144881. Epub 2016 Feb 18. PMID 26892479
- [Background] Fielding AK, Rowe JM, Buck G, Foroni L, Gerrard G, Litzow MR, Lazarus H, Luger SM, Marks DI, McMillan AK, Moorman AV, Patel B, Paietta E, Tallman MS, Goldstone AH. UKALLXII/ECOG2993: addition of imatinib to a standard treatment regimen enhances long-term outcomes in Philadelphia positive acute lymphoblastic leukemia. Blood. 2014 Feb 6;123(6):843-50. doi: 10.1182/blood-2013-09-529008. Epub 2013 Nov 25. PMID 24277073
- [Background] Fielding AK, Rowe JM, Richards SM, Buck G, Moorman AV, Durrant IJ, Marks DI, McMillan AK, Litzow MR, Lazarus HM, Foroni L, Dewald G, Franklin IM, Luger SM, Paietta E, Wiernik PH, Tallman MS, Goldstone AH. Prospective outcome data on 267 unselected adult patients with Philadelphia chromosome-positive acute lymphoblastic leukemia confirms superiority of allogeneic transplantation over chemotherapy in the pre-imatinib era: results from the International ALL Trial MRC UKALLXII/ECOG2993. Blood. 2009 May 7;113(19):4489-96. doi: 10.1182/blood-2009-01-199380. Epub 2009 Feb 24. PMID 19244158
- [Background] Foa R, Vitale A, Vignetti M, Meloni G, Guarini A, De Propris MS, Elia L, Paoloni F, Fazi P, Cimino G, Nobile F, Ferrara F, Castagnola C, Sica S, Leoni P, Zuffa E, Fozza C, Luppi M, Candoni A, Iacobucci I, Soverini S, Mandelli F, Martinelli G, Baccarani M; GIMEMA Acute Leukemia Working Party. Dasatinib as first-line treatment for adult patients with Philadelphia chromosome-positive acute lymphoblastic leukemia. Blood. 2011 Dec 15;118(25):6521-8. doi: 10.1182/blood-2011-05-351403. Epub 2011 Sep 19. PMID 21931113
- [Background] Chiaretti S, Vitale A, Vignetti M, Piciocchi A, Fazi P, Elia L, Falini B, Ronco F, Ferrara F, De Fabritiis P, Luppi M, La Nasa G, Tedeschi A, Califano C, Fanin R, Dore F, Mandelli F, Meloni G, Foa R. A sequential approach with imatinib, chemotherapy and transplant for adult Ph+ acute lymphoblastic leukemia: final results of the GIMEMA LAL 0904 study. Haematologica. 2016 Dec;101(12):1544-1552. doi: 10.3324/haematol.2016.144535. Epub 2016 Aug 11. PMID 27515250
- [Background] Kantarjian H, Giles F, Wunderle L, Bhalla K, O'Brien S, Wassmann B, Tanaka C, Manley P, Rae P, Mietlowski W, Bochinski K, Hochhaus A, Griffin JD, Hoelzer D, Albitar M, Dugan M, Cortes J, Alland L, Ottmann OG. Nilotinib in imatinib-resistant CML and Philadelphia chromosome-positive ALL. N Engl J Med. 2006 Jun 15;354(24):2542-51. doi: 10.1056/NEJMoa055104. PMID 16775235
- [Background] Kim DY, Joo YD, Lim SN, Kim SD, Lee JH, Lee JH, Kim DH, Kim K, Jung CW, Kim I, Yoon SS, Park S, Ahn JS, Yang DH, Lee JJ, Lee HS, Kim YS, Mun YC, Kim H, Park JH, Moon JH, Sohn SK, Lee SM, Lee WS, Kim KH, Won JH, Hyun MS, Park J, Lee JH, Shin HJ, Chung JS, Lee H, Eom HS, Lee GW, Cho YU, Jang S, Park CJ, Chi HS, Lee KH; Adult Acute Lymphoblastic Leukemia Working Party of the Korean Society of Hematology. Nilotinib combined with multiagent chemotherapy for newly diagnosed Philadelphia-positive acute lymphoblastic leukemia. Blood. 2015 Aug 6;126(6):746-56. doi: 10.1182/blood-2015-03-636548. Epub 2015 Jun 11. PMID 26065651
- [Background] Laport GG, Alvarnas JC, Palmer JM, Snyder DS, Slovak ML, Cherry AM, Wong RM, Negrin RS, Blume KG, Forman SJ. Long-term remission of Philadelphia chromosome-positive acute lymphoblastic leukemia after allogeneic hematopoietic cell transplantation from matched sibling donors: a 20-year experience with the fractionated total body irradiation-etoposide regimen. Blood. 2008 Aug 1;112(3):903-9. doi: 10.1182/blood-2008-03-143115. Epub 2008 Jun 2. PMID 18519812
- [Background] Lee KH, Lee JH, Choi SJ, Lee JH, Seol M, Lee YS, Kim WK, Lee JS, Seo EJ, Jang S, Park CJ, Chi HS. Clinical effect of imatinib added to intensive combination chemotherapy for newly diagnosed Philadelphia chromosome-positive acute lymphoblastic leukemia. Leukemia. 2005 Sep;19(9):1509-16. doi: 10.1038/sj.leu.2403886. PMID 16034462
- [Background] Machova Polakova K, Kulvait V, Benesova A, Linhartova J, Klamova H, Jaruskova M, de Benedittis C, Haferlach T, Baccarani M, Martinelli G, Stopka T, Ernst T, Hochhaus A, Kohlmann A, Soverini S. Next-generation deep sequencing improves detection of BCR-ABL1 kinase domain mutations emerging under tyrosine kinase inhibitor treatment of chronic myeloid leukemia patients in chronic phase. J Cancer Res Clin Oncol. 2015 May;141(5):887-99. doi: 10.1007/s00432-014-1845-6. Epub 2014 Nov 4. PMID 25367136
- [Background] Mastrangelo R, Poplack D, Bleyer A, Riccardi R, Sather H, D'Angio G. Report and recommendations of the Rome workshop concerning poor-prognosis acute lymphoblastic leukemia in children: biologic bases for staging, stratification, and treatment. Med Pediatr Oncol. 1986;14(3):191-4. doi: 10.1002/mpo.2950140317. No abstract available. PMID 3528788
- [Background] Mizuta S, Matsuo K, Nishiwaki S, Imai K, Kanamori H, Ohashi K, Fukuda T, Onishi Y, Miyamura K, Takahashi S, Onizuka M, Atsuta Y, Suzuki R, Morishima Y, Kato K, Sakamaki H, Tanaka J. Pretransplant administration of imatinib for allo-HSCT in patients with BCR-ABL-positive acute lymphoblastic leukemia. Blood. 2014 Apr 10;123(15):2325-32. doi: 10.1182/blood-2013-11-538728. Epub 2014 Mar 3. PMID 24591204
- [Background] Ottmann O, Dombret H, Martinelli G, Simonsson B, Guilhot F, Larson RA, Rege-Cambrin G, Radich J, Hochhaus A, Apanovitch AM, Gollerkeri A, Coutre S. Dasatinib induces rapid hematologic and cytogenetic responses in adult patients with Philadelphia chromosome positive acute lymphoblastic leukemia with resistance or intolerance to imatinib: interim results of a phase 2 study. Blood. 2007 Oct 1;110(7):2309-15. doi: 10.1182/blood-2007-02-073528. Epub 2007 May 11. PMID 17496201
- [Background] Ravandi F. Current management of Philadelphia chromosome positive ALL and the role of stem cell transplantation. Hematology Am Soc Hematol Educ Program. 2017 Dec 8;2017(1):22-27. doi: 10.1182/asheducation-2017.1.22. PMID 29222233
- [Background] Ravandi F, Jorgensen JL, Thomas DA, O'Brien S, Garris R, Faderl S, Huang X, Wen S, Burger JA, Ferrajoli A, Kebriaei P, Champlin RE, Estrov Z, Challagundla P, Wang SA, Luthra R, Cortes JE, Kantarjian HM. Detection of MRD may predict the outcome of patients with Philadelphia chromosome-positive ALL treated with tyrosine kinase inhibitors plus chemotherapy. Blood. 2013 Aug 15;122(7):1214-21. doi: 10.1182/blood-2012-11-466482. Epub 2013 Jul 8. PMID 23836561
- [Background] Ravandi F, O'Brien S, Thomas D, Faderl S, Jones D, Garris R, Dara S, Jorgensen J, Kebriaei P, Champlin R, Borthakur G, Burger J, Ferrajoli A, Garcia-Manero G, Wierda W, Cortes J, Kantarjian H. First report of phase 2 study of dasatinib with hyper-CVAD for the frontline treatment of patients with Philadelphia chromosome-positive (Ph+) acute lymphoblastic leukemia. Blood. 2010 Sep 23;116(12):2070-7. doi: 10.1182/blood-2009-12-261586. Epub 2010 May 13. PMID 20466853
- [Background] Ravandi F, O'Brien SM, Cortes JE, Thomas DM, Garris R, Faderl S, Burger JA, Rytting ME, Ferrajoli A, Wierda WG, Verstovsek S, Champlin R, Kebriaei P, McCue DA, Huang X, Jabbour E, Garcia-Manero G, Estrov Z, Kantarjian HM. Long-term follow-up of a phase 2 study of chemotherapy plus dasatinib for the initial treatment of patients with Philadelphia chromosome-positive acute lymphoblastic leukemia. Cancer. 2015 Dec 1;121(23):4158-64. doi: 10.1002/cncr.29646. Epub 2015 Aug 26. PMID 26308885
- [Background] Ravandi F, Othus M, O'Brien SM, Forman SJ, Ha CS, Wong JYC, Tallman MS, Paietta E, Racevskis J, Uy GL, Horowitz M, Takebe N, Little R, Borate U, Kebriaei P, Kingsbury L, Kantarjian HM, Radich JP, Erba HP, Appelbaum FR. US Intergroup Study of Chemotherapy Plus Dasatinib and Allogeneic Stem Cell Transplant in Philadelphia Chromosome Positive ALL. Blood Adv. 2016 Dec 27;1(3):250-259. doi: 10.1182/bloodadvances.2016001495. PMID 29046900
- [Background] Rousselot P, Coude MM, Gokbuget N, Gambacorti Passerini C, Hayette S, Cayuela JM, Huguet F, Leguay T, Chevallier P, Salanoubat C, Bonmati C, Alexis M, Hunault M, Glaisner S, Agape P, Berthou C, Jourdan E, Fernandes J, Sutton L, Banos A, Reman O, Lioure B, Thomas X, Ifrah N, Lafage-Pochitaloff M, Bornand A, Morisset L, Robin V, Pfeifer H, Delannoy A, Ribera J, Bassan R, Delord M, Hoelzer D, Dombret H, Ottmann OG; European Working Group on Adult ALL (EWALL) group. Dasatinib and low-intensity chemotherapy in elderly patients with Philadelphia chromosome-positive ALL. Blood. 2016 Aug 11;128(6):774-82. doi: 10.1182/blood-2016-02-700153. Epub 2016 Apr 27. PMID 27121472
- [Background] Salek C, Folber F, Fronkova E, Prochazka B, Marinov I, Cetkovsky P, Mayer J, Doubek M; Czech Leukemia Study Group - for Life. Early MRD response as a prognostic factor in adult patients with acute lymphoblastic leukemia. Eur J Haematol. 2016 Mar;96(3):276-84. doi: 10.1111/ejh.12587. Epub 2015 Jun 22. PMID 25997106
- [Background] Short NJ, Jabbour E, Sasaki K, Patel K, O'Brien SM, Cortes JE, Garris R, Issa GC, Garcia-Manero G, Luthra R, Thomas D, Kantarjian H, Ravandi F. Impact of complete molecular response on survival in patients with Philadelphia chromosome-positive acute lymphoblastic leukemia. Blood. 2016 Jul 28;128(4):504-7. doi: 10.1182/blood-2016-03-707562. Epub 2016 May 27. PMID 27235138
- [Background] Schultz KR, Bowman WP, Aledo A, Slayton WB, Sather H, Devidas M, Wang C, Davies SM, Gaynon PS, Trigg M, Rutledge R, Burden L, Jorstad D, Carroll A, Heerema NA, Winick N, Borowitz MJ, Hunger SP, Carroll WL, Camitta B. Improved early event-free survival with imatinib in Philadelphia chromosome-positive acute lymphoblastic leukemia: a children's oncology group study. J Clin Oncol. 2009 Nov 1;27(31):5175-81. doi: 10.1200/JCO.2008.21.2514. Epub 2009 Oct 5. PMID 19805687
- [Background] Tanguy-Schmidt A, Rousselot P, Chalandon Y, Cayuela JM, Hayette S, Vekemans MC, Escoffre M, Huguet F, Rea D, Delannoy A, Cahn JY, Vernant JP, Ifrah N, Dombret H, Thomas X. Long-term follow-up of the imatinib GRAAPH-2003 study in newly diagnosed patients with de novo Philadelphia chromosome-positive acute lymphoblastic leukemia: a GRAALL study. Biol Blood Marrow Transplant. 2013 Jan;19(1):150-5. doi: 10.1016/j.bbmt.2012.08.021. Epub 2012 Sep 6. PMID 22960387
- [Background] Vignetti M, Fazi P, Cimino G, Martinelli G, Di Raimondo F, Ferrara F, Meloni G, Ambrosetti A, Quarta G, Pagano L, Rege-Cambrin G, Elia L, Bertieri R, Annino L, Foa R, Baccarani M, Mandelli F. Imatinib plus steroids induces complete remissions and prolonged survival in elderly Philadelphia chromosome-positive patients with acute lymphoblastic leukemia without additional chemotherapy: results of the Gruppo Italiano Malattie Ematologiche dell'Adulto (GIMEMA) LAL0201-B protocol. Blood. 2007 May 1;109(9):3676-8. doi: 10.1182/blood-2006-10-052746. Epub 2007 Jan 9. PMID 17213285
- [Background] Wetzler M, Watson D, Stock W, Koval G, Mulkey FA, Hoke EE, McCarty JM, Blum WG, Powell BL, Marcucci G, Bloomfield CD, Linker CA, Larson RA. Autologous transplantation for Philadelphia chromosome-positive acute lymphoblastic leukemia achieves outcomes similar to allogeneic transplantation: results of CALGB Study 10001 (Alliance). Haematologica. 2014 Jan;99(1):111-5. doi: 10.3324/haematol.2013.085811. Epub 2013 Sep 27. PMID 24077846
- [Background] Yanada M, Takeuchi J, Sugiura I, Akiyama H, Usui N, Yagasaki F, Kobayashi T, Ueda Y, Takeuchi M, Miyawaki S, Maruta A, Emi N, Miyazaki Y, Ohtake S, Jinnai I, Matsuo K, Naoe T, Ohno R; Japan Adult Leukemia Study Group. High complete remission rate and promising outcome by combination of imatinib and chemotherapy for newly diagnosed BCR-ABL-positive acute lymphoblastic leukemia: a phase II study by the Japan Adult Leukemia Study Group. J Clin Oncol. 2006 Jan 20;24(3):460-6. doi: 10.1200/JCO.2005.03.2177. Epub 2005 Dec 12. PMID 16344315
- [Result] Chalandon Y, Thomas X, Hayette S, Cayuela JM, Abbal C, Huguet F, Raffoux E, Leguay T, Rousselot P, Lepretre S, Escoffre-Barbe M, Maury S, Berthon C, Tavernier E, Lambert JF, Lafage-Pochitaloff M, Lheritier V, Chevret S, Ifrah N, Dombret H; Group for Research on Adult Acute Lymphoblastic Leukemia (GRAALL). Randomized study of reduced-intensity chemotherapy combined with imatinib in adults with Ph-positive acute lymphoblastic leukemia. Blood. 2015 Jun 11;125(24):3711-9. doi: 10.1182/blood-2015-02-627935. Epub 2015 Apr 15. PMID 25878120
- [Result] Dorer DJ, Knickerbocker RK, Baccarani M, Cortes JE, Hochhaus A, Talpaz M, Haluska FG. Impact of dose intensity of ponatinib on selected adverse events: Multivariate analyses from a pooled population of clinical trial patients. Leuk Res. 2016 Sep;48:84-91. doi: 10.1016/j.leukres.2016.07.007. Epub 2016 Jul 22. PMID 27505637
- [Result] Jabbour E, Kantarjian H, Ravandi F, Thomas D, Huang X, Faderl S, Pemmaraju N, Daver N, Garcia-Manero G, Sasaki K, Cortes J, Garris R, Yin CC, Khoury JD, Jorgensen J, Estrov Z, Bohannan Z, Konopleva M, Kadia T, Jain N, DiNardo C, Wierda W, Jeanis V, O'Brien S. Combination of hyper-CVAD with ponatinib as first-line therapy for patients with Philadelphia chromosome-positive acute lymphoblastic leukaemia: a single-centre, phase 2 study. Lancet Oncol. 2015 Nov;16(15):1547-1555. doi: 10.1016/S1470-2045(15)00207-7. Epub 2015 Sep 30. PMID 26432046
- See also: Acute Lymphocytic Leukemia — https://vsearch.nlm.nih.gov/vivisimo/cgi-bin/query-meta?v%3aproject=medlineplus&v%3asources=medlineplus-bundle&query=Acute%20lymphocytic%20Leukemia&
- See also: Ponatinib — https://druginfo.nlm.nih.gov/drugportal/name/Ponatinib+hydrochloride